CLINICAL TRIAL: NCT06890169
Title: OneSTOP (One-Stop Telehealth Obesity Program): the Use of Telecare and Digital Platforms for Multidisciplinary Management of Weight Management and Related Comorbidities
Brief Title: OneSTOP (One-Stop Telehealth Obesity Program) for Multidisciplinary Weight Management and Related Comorbidities
Acronym: OneSTOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Joan Khoo Joo Ching, Clinical Associate Professor, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OneSTOP Empower
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Type 2 Diabetes; NAFLD - Non-Alcoholic Fatty Liver Disease; Hypertension; Dyslipidaemia; Telemedicine
Keywords: obesity; type 2 diabetes; masld; nafld; telecare; telemedicine
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The standard F2F structured weight management program consists of 4 doctor and 4 dietician consults over 26 weeks, at 2-4 weekly intervals in the first 3 months, and 6-8 weeks in the next 3 months. At the baseline visit, participants are provided with an aerobic and resistance exercise prescription individualized to each subject's fitness and comorbidities to target at least 180 minutes/week of moderate-intensity physical activity (with exercise on at least 3 days/week), and dietary advice based on a calorie-deficit diet (400-600 kilocalories less than the calculated daily caloric requirement, based on the Mifflin-St Jeor equation) which emphasizes reduction in sugar-sweetened beverages, refined carbohydrates and saturated fats. Subjects will be provided with a list of fitness resources such as gyms and fitness corners with advice on use of the equipment, and specific guidance on increasing intensity and duration of exercise and monitoring for injury.
  Interventions: Behavioral: Standard of care weight management program
- OneSTOP program (Experimental): The OneSTOP program will incorporate at least 50% (4 out of 8 sessions) of the doctor and dietician consults over the 26-week study as teleconsults, which may be scheduled as joint or asynchronous consults. The exercise prescription and calorie restriction will be tailored to each subject's individual needs as in the F2F structured weight management program in the control group. In addition, participants will be taught to use the EMPOWER app will be used to enable them to upload their weight, blood pressure and glucose, food and exercise duration records. The app also has the capability to co-ordinate visits and investigations, deliver intelligent health nudges and reminders on adherence to treatment which can be individualized to their progress, and provide information on their conditions curated by their doctors and dieticians.
  Interventions: Behavioral: OneSTOP program

INTERVENTIONS:
Behavioral: OneSTOP program — The OneSTOP program will incorporate at least 50% (4 out of 8 sessions) of the doctor and dietician consults over the 26-week study as teleconsults, which may be scheduled as joint or asynchronous consults. The exercise prescription and calorie restriction will be tailored to each subject's individual needs as in the F2F structured weight management program in the control group. In addition, participants will be taught to use the EMPOWER app will be used to enable them to upload their weight, blood pressure and glucose, food and exercise duration records. The app also has the capability to co-ordinate visits and investigations, deliver intelligent health nudges and reminders on adherence to treatment which can be individualized to their progress, and provide information on their conditions curated by their doctors and dieticians.
  Arms: OneSTOP program
Behavioral: Standard of care weight management program — The standard face-to-face weight management program consists of 4 doctor and 4 dietician consults over 26 weeks, at 2-4 weekly intervals in the first 3 months, and 6-8 weeks in the next 3 months. At the baseline visit, participants are provided with an aerobic and resistance exercise prescription individualized to each subject's fitness and comorbidities to target at least 180 minutes/week of moderate-intensity physical activity (with exercise on at least 3 days/week), and dietary advice based on a calorie-deficit diet (400-600 kilocalories less than the calculated daily caloric requirement, based on the Mifflin-St Jeor equation) which emphasizes reduction in sugar-sweetened beverages, refined carbohydrates and saturated fats. Subjects will be provided with a list of fitness resources such as gyms and fitness corners with advice on use of the equipment, and specific guidance on increasing intensity and duration of exercise and monitoring for injury.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if the use of a care model including teleconsults and the EMPOWER app can induce clinically significant weight loss and metabolic improvements in obese adults with diabetes and metabolic dysfunction-associated steatotic liver disease (MASLD).

Researchers will compare this model with the conventional standard of care of physical visit-based weight management program to see if this model is non-inferior to the standard of care for inducing weight loss, and if there is greater patient convenience with telehealth and more frequent self-monitoring, compliance with diet advice and exercise participation compared to standard of care.

Participants in the standard arm will attend 4 physical doctor and 4 physical dietician consultations over 26 weeks, where they will be provided with an individualized diet and exercise prescription to induce at least 5% weight loss.

Participants in the intervention arm will have the same number of consults over 26 weeks, of which at least 50% will be teleconsults, and will also be provided with an individualized diet and exercise prescription to induce at least 5% weight loss. In addition, they will be taught to use the EMPOWER app to upload weight, blood pressure and glucose, food and exercise records which will be reviewed at the consults. The app also delivers nudges to improve adherence to lifestyle modification.

DETAILED DESCRIPTION:
Design This a randomized controlled study comparing a standard weight management program of face-to-face (F2F) consults with doctors (endocrinologists and sports medicine physicians) and dieticians as defined by best-practice guidelines (control), or to the OneSTOP (One-Stop Telecare Obesity Program) a novel weight management intervention incorporating telecare and the EMPOWER app jointly developed by SingHealth and the NUS School of Computing.

Standard of care (control) The standard F2F structured weight management program consists of 4 doctor and 4 dietician consults over 26 weeks, at 2-4 weekly intervals in the first 3 months, and 6-8 weeks in the next 3 months. At the baseline visit, participants are provided with an aerobic and resistance exercise prescription individualized to each subject's fitness and comorbidities to target at least 180 minutes/week of moderate-intensity physical activity (with exercise on at least 3 days/week), and dietary advice based on a calorie-deficit diet (400-600 kilocalories less than the calculated daily caloric requirement, based on the Mifflin-St Jeor equation) which emphasizes reduction in sugar-sweetened beverages, refined carbohydrates and saturated fats. Subjects will be provided with a list of fitness resources such as gyms and fitness corners with advice on use of the equipment, and specific guidance on increasing intensity and duration of exercise and monitoring for injury. Dietary advice will be based on standard guidelines to target a calorie-deficit of 400-600 kcal from baseline. All subjects will keep food diaries and records of exercise duration for review and will also be provided with links to online resources for health advice and generic apps to track their calorie intake and physical activity. At each visit, exercise and diet records and/or results of investigations will be reviewed, and lifestyle advice modified to target at least 5% weight loss.

Intervention This will incorporate at least 50% (4 out of 8 sessions) of the doctor and dietician consults over the 26-week study as teleconsults, which may be scheduled as joint or asynchronous consults. The exercise prescription will likewise be tailored to each subject's individual needs as in the F2F structured weight management program in the control group, and similar dietary advice and reviews will be provided. In addition, participants will be taught to use the EMPOWER app will be used to enable them to upload their weight, blood pressure and glucose, food and exercise duration records. The app also has the capability to co-ordinate visits and investigations, deliver intelligent health nudges and reminders on adherence to treatment which can be individualized to their progress, and provide information on their conditions with additional information curated by their doctors and dieticians. Subjects will be able to compare the photos of their food with that in a database on the app, which will make calorie counting more precise. The app will also be paired with an activity tracker for more accurate estimates of exercise duration. Similar to the standard program, doctors and dieticians will review the exercise and diet records, results of investigations, and modify treatment according to patient response, according to standard care guidelines, aiming for at least 5% weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-70
* Body mass index > 27.5 kg/m2
* Waist circumference > 90 cm in men or 80 cm in women
* Suboptimal control of type 2 diabetes (HbA1c > 6.5%) AND/OR MASLD (as defined on radiological or histological evidence of hepatic steatosis in the absence of other chronic liver disease)

Exclusion Criteria:

* Men who drink > 21 units/week and women who drink > 14 units/week of alcohol
* Participants previously on weight-lowering medications (however if they are keen to participate, there will be a minimum wash-out period of 3 months before participation)
* Illness with life expectancy of less than 6 months
* Inability to comply with written instructions in English

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
weight loss | 26 weeks
  percentage reduction in weight from baseline

SECONDARY OUTCOMES:
percentage of subjects with reduction in weight at least 5% | 26 weeks
  percentage of subjects with reduction in weight at least 5%
improvement in glycaemic control | 26 weeks
  reduction in HbA1c
improvement in MASLD | 26 weeks
  reduction in severity of MASLD using liver function tests and imaging to measure hepatic steatosis and fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, MBBS, FRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Data of patients is confidential.